CLINICAL TRIAL: NCT04744675
Title: Peripheral Nerve Injections for the Treatment of Upper Extremity Complex Regional Pain Syndrome: a Feasibility Study for a Proposed Randomized Design
Brief Title: Peripheral Nerve Injections for CRPS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20200600-01H
Record Dates: First submitted 2021-01-21; First posted 2021-02-09 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Complex Regional Pain Syndromes
MeSH Terms: conditions — Complex Regional Pain Syndromes | interventions — Triamcinolone Acetonide; Sodium Chloride; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): The intervention group will receive:
  1. Suprascapular nerve block - 3 mL of 0.5% Bupivacaine and 1 mL of 40 mg/mL Kenalog
  2. Median nerve block - 3.5 mL of 0.5% Bupivacaine and 0.5 mL of 40 mg/mL Kenalog
  3. Ulnar nerve block - 3.5 mL of 0.5% Bupivacaine and 0.5 mL of 40 mg/mL Kenalog
  Interventions: Drug: Triamcinolone Acetonide 40mg/mL; Drug: Bupivacaine
- Placebo (Placebo Comparator): Placebo
  The placebo group will receive:
  1. Suprascapular nerve injection - 4 mL of normal saline
  2. Median nerve injection - 4 mL of normal saline
  3. Ulnar nerve injection - 4 mL of normal saline
  Interventions: Drug: Saline Injection

INTERVENTIONS:
Drug: Triamcinolone Acetonide 40mg/mL — Triamcinolone acetonide is a synthetic glucocorticoid corticosteroid with marked anti-inflammatory action, in a sterile aqueous suspension suitable for intramuscular, intra-articular, and intrabursal injection.
  Other Names: Kenalog
  Arms: Treatment
Drug: Saline Injection — Saline is a buffer solution commonly used in biological research. It is a water-based salt solution containing disodium hydrogen phosphate, sodium chloride and, in some formulations, potassium chloride and potassium dihydrogen phosphate. The buffer helps to maintain a constant pH. The osmolarity and ion concentrations of the solutions match those of the human body.
  Arms: Placebo
Drug: Bupivacaine — Bupivacaine is an anesthetic that is commonly used as a local numbing agent, including intramuscular, intra-articular and intrabursal injections.
  Other Names: Marcaine
  Arms: Treatment

SUMMARY:
Background Complex regional pain syndrome (CRPS) is characterized by intense pain, loss of function, and associated with motor, trophic, sudomotor, and/or vasomotor changes of the affected extremity. Upper extremity CRPS is seen frequently in electrodiagnostic, neurology, and musculoskeletal clinics and occurs in up to one-third of patients who have undergone common surgical procedures (i.e. carpal tunnel surgery). To date, there is a limited understanding of the underlying pathophysiology of CRPS. As a consequence, few effective treatment options are available.

Peripheral nerve blocks have proven to be successful in reducing pain for several musculoskeletal and neurologic conditions. Similarly, this procedure could be used to block somatic and autonomic sensory fibers which are thought to contribute to CRPS. In a small exploratory study, investigators found peripheral nerve blocks in the upper extremity (suprascapular and median nerves) were well-tolerated in patients with CRPS and resulted in a 56% and 37% pain reduction in the shoulder and hand 2 weeks after injection, respectively. While this is highly encouraging, large randomized placebo-controlled trials (RCTs) are necessary to demonstrate effectiveness and safety of nerve blocks for this population before it is accepted into clinical practice. This proposal is a phase II feasibility study that will test the critical elements necessary for performing such a RCT.

Methods The investigators will recruit participants (≥18 years old) from The Ottawa Hospital, Bruyère Continuing Care (Elisabeth Bruyère Hospital, St-Vincent Hospital), and Providence Care Hospital (Kingston, ON), meeting the well-established clinical Budapest criteria for upper extremity CRPS and having a visual analog scale (VAS) pain score of at least 40 mm (to avoid flooring effect). Participants will be block-randomized by the Ottawa Methods Centre to receive injections of either A) intervention (suprascapular, median, and ulnar nerves) with bupivacaine and triamcinolone acetonide, or B) placebo (saline). All participants will receive standard care for CRPS.

Primary outcomes will focus on crucial methodologic aspects for the future RCT, including: (1) level of recruitment, (2) rate of acceptance from eligible patients to the randomization procedure, (3) blinding efficacy, (4) degree of patient retention, (5) rate of data completion, and (6) rate of adverse events for both the placebo and intervention groups.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide signed and dated informed consent form
2. Male or female, aged ≥18 years old
3. Satisfy the Budapest Criteria for upper extremity CRPS
4. A VAS score of at least 40 mm in the upper extremity to avoid flooring effect for injection-related pain reduction

Exclusion Criteria:

1. Uncontrolled hypertension (>180/110)
2. Sepsis
3. Bleeding diathesis
4. Active cancer
5. Brachial plexus injuries
6. Neurological language deficits precluding participation
7. Mini mental state examination score < 23
8. Acute mental illness (An acute mental illness is characterized by clinically significant symptoms of any metal health illness that requires immediate treatment. The physician making the recommendation to be part of the study. If the patient exhibits symptoms of any mental health illness that is not being treated by either the recommending physician or another member of the patient's care team the patient will not be recommended to participate in the study)
9. Patients who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Recruitment | Week -2
  Number of participants who are successfully recruit into the study.
Randomization | Week 0
  Number of participants who accept being randomized into either the intervention or placebo treatment arms and receive the injection accordingly.
Blinding - Participant | Week 0
  The participants will be asked which arm they believe they are part of and this response will be compared to their actual group allocation. The level of agreement between the actual group allocation and the guess provided will be compared using Bang's blinding index, we will consider blinding effective if the index is between -0.2 and 0.2 (zero being perfect blinding).
Blinding - Participant | Week 2
  The participants will be asked which arm they believe they are part of and this response will be compared to their actual group allocation. The level of agreement between the actual group allocation and the guess provided will be compared using Bang's blinding index, we will consider blinding effective if the index is between -0.2 and 0.2 (zero being perfect blinding).
Blinding - Participant | Week 6
  The participants will be asked which arm they believe they are part of and this response will be compared to their actual group allocation. The level of agreement between the actual group allocation and the guess provided will be compared using Bang's blinding index, we will consider blinding effective if the index is between -0.2 and 0.2 (zero being perfect blinding).
Blinding - Participant | Week 12
  The participants will be asked which arm they believe they are part of and this response will be compared to their actual group allocation. The level of agreement between the actual group allocation and the guess provided will be compared using Bang's blinding index, we will consider blinding effective if the index is between -0.2 and 0.2 (zero being perfect blinding).
Blinding - Interventionist | Week 0
  The interventionist will be asked which arm they believe the participant is are part of and this response will be compared to their actual group allocation. The level of agreement between the actual group allocation and the guess provided will be compared using Bang's blinding index, we will consider blinding effective if the index is between -0.2 and 0.2 (zero being perfect blinding).
Blinding - Physiotherapist | Week 2
  The physiotherapist will be asked which arm they believe the participant is are part of and this response will be compared to their actual group allocation. The level of agreement between the actual group allocation and the guess provided will be compared using Bang's blinding index, we will consider blinding effective if the index is between -0.2 and 0.2 (zero being perfect blinding).
Blinding - Physiotherapist | Week 6
  The physiotherapist will be asked which arm they believe the participant is are part of and this response will be compared to their actual group allocation. The level of agreement between the actual group allocation and the guess provided will be compared using Bang's blinding index, we will consider blinding effective if the index is between -0.2 and 0.2 (zero being perfect blinding).
Blinding - Physiotherapist | Week 12
  The physiotherapist will be asked which arm they believe the participant is are part of and this response will be compared to their actual group allocation. The level of agreement between the actual group allocation and the guess provided will be compared using Bang's blinding index, we will consider blinding effective if the index is between -0.2 and 0.2 (zero being perfect blinding).
Retention | Week 12
  The percentage of participants who remained in the study for the entire duration of their planned involvement.
Data completion | Week 12
  The percentage of participants who complete all of the study questionnaires
Rate of Adverse events | Week 12
  We will track adverse events the participants experience

SECONDARY OUTCOMES:
Pain - Visual Analog Scale | Week -2
  We will track the pain experienced by the participants on a visual analog scale. The lowest score is 0 the highest score is 10. A higher value indicates a higher amount of pain experienced by the participant
Pain - Visual Analog Scale | Week 0 - Immediately before injection
  We will track the pain experienced by the participants on a visual analog scale. The lowest score is 0 the highest score is 10. A higher value indicates a higher amount of pain experienced by the participant
Pain - Visual Analog Scale | Week 0 - Immediately after injection
  We will track the pain experienced by the participants on a visual analog scale. The lowest score is 0 the highest score is 10. A higher value indicates a higher amount of pain experienced by the participant
Pain - Visual Analog Scale | Week 2
  We will track the pain experienced by the participants on a visual analog scale. The lowest score is 0 the highest score is 10. A higher value indicates a higher amount of pain experienced by the participant
Pain - Visual Analog Scale | Week 6
  We will track the pain experienced by the participants on a visual analog scale. The lowest score is 0 the highest score is 10. A higher value indicates a higher amount of pain experienced by the participant
Pain - Visual Analog Scale | Week 12
  We will track the pain experienced by the participants on a visual analog scale. The lowest score is 0 the highest score is 10. A higher value indicates a higher amount of pain experienced by the participant
Pain - Patient-Reported Outcomes Measurement Information System 29 Profile V2 | Week -2
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 4 and the highest possible score is 30, and a higher score indicates a worse outcome.
Pain - Patient-Reported Outcomes Measurement Information System 29 Profile V2 | Week 0
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 4 and the highest possible score is 30, and a higher score indicates a worse outcome.
Pain - Patient-Reported Outcomes Measurement Information System 29 Profile V2 | Week 2
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 4 and the highest possible score is 30, and a higher score indicates a worse outcome.
Pain - Patient-Reported Outcomes Measurement Information System 29 Profile V2 | Week 6
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 4 and the highest possible score is 30, and a higher score indicates a worse outcome.
Pain - Patient-Reported Outcomes Measurement Information System 29 Profile V2 | Week 12
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 4 and the highest possible score is 30, and a higher score indicates a worse outcome.
Pain - EQ-5D-5L | Week -2
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 1 and the highest possible score is 5, and a higher score indicates a worse outcome.
Pain - EQ-5D-5L | Week 0
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 1 and the highest possible score is 5, and a higher score indicates a worse outcome.
Pain - EQ-5D-5L | Week 2
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 1 and the highest possible score is 5, and a higher score indicates a worse outcome.
Pain - EQ-5D-5L | Week 6
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 1 and the highest possible score is 5, and a higher score indicates a worse outcome.
Pain - EQ-5D-5L | Week 12
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 1 and the highest possible score is 5, and a higher score indicates a worse outcome.
Disease Severity - Complex Regional Pain Syndrome Severity Score | Week -2
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 0 and the highest possible score is 17, and a higher score indicates a worse outcome.
Disease Severity - Complex Regional Pain Syndrome Severity Score | Week 0
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 0 and the highest possible score is 17, and a higher score indicates a worse outcome.
Disease Severity - Complex Regional Pain Syndrome Severity Score | Week 2
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 0 and the highest possible score is 17, and a higher score indicates a worse outcome.
Disease Severity - Complex Regional Pain Syndrome Severity Score | Week 6
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 0 and the highest possible score is 17, and a higher score indicates a worse outcome.
Disease Severity - Complex Regional Pain Syndrome Severity Score | Week 12
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 0 and the highest possible score is 17, and a higher score indicates a worse outcome.
Function - Disabilities of the Arm, Shoulder, and Hand Questionnaire | Week -2
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 0 and the highest possible score is 100, and a higher score indicates a worse outcome.
Function - Disabilities of the Arm, Shoulder, and Hand Questionnaire | Week 0
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 0 and the highest possible score is 100, and a higher score indicates a worse outcome.
Function - Disabilities of the Arm, Shoulder, and Hand Questionnaire | Week 2
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 0 and the highest possible score is 100, and a higher score indicates a worse outcome.
Function - Disabilities of the Arm, Shoulder, and Hand Questionnaire | Week 6
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 0 and the highest possible score is 100, and a higher score indicates a worse outcome.
Function - Disabilities of the Arm, Shoulder, and Hand Questionnaire | Week 12
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 0 and the highest possible score is 100, and a higher score indicates a worse outcome.
Function - Patient-Reported Outcomes Measurement Information System 29 Profile V2 | Week -2
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 8 and the highest possible score is 40, and a higher score indicates a better outcome.
Function - Patient-Reported Outcomes Measurement Information System 29 Profile V2 | Week 0
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 8 and the highest possible score is 40, and a higher score indicates a better outcome.
Function - Patient-Reported Outcomes Measurement Information System 29 Profile V2 | Week 2
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 8 and the highest possible score is 40, and a higher score indicates a better outcome.
Function - Patient-Reported Outcomes Measurement Information System 29 Profile V2 | Week 6
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 8 and the highest possible score is 40, and a higher score indicates a better outcome.
Function - Patient-Reported Outcomes Measurement Information System 29 Profile V2 | Week 12
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 8 and the highest possible score is 40, and a higher score indicates a better outcome.
Emotional and Psychological Function - Patient-Reported Outcomes Measurement Information System 29 Profile V2 | Week -2
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 16 and the highest possible score is 80, and a higher score indicates a worse outcome.
Emotional and Psychological Function - Patient-Reported Outcomes Measurement Information System 29 Profile V2 | Week 0
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 16 and the highest possible score is 80, and a higher score indicates a worse outcome.
Emotional and Psychological Function - Patient-Reported Outcomes Measurement Information System 29 Profile V2 | Week 2
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 16 and the highest possible score is 80, and a higher score indicates a worse outcome.
Emotional and Psychological Function - Patient-Reported Outcomes Measurement Information System 29 Profile V2 | Week 6
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 16 and the highest possible score is 80, and a higher score indicates a worse outcome.
Emotional and Psychological Function - Patient-Reported Outcomes Measurement Information System 29 Profile V2 | Week 12
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 16 and the highest possible score is 80, and a higher score indicates a worse outcome.
Emotional and Psychological Function - EQ-5D-5L | Week -2
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 1 and the highest possible score is 5, and a higher score indicates a worse outcome.
Emotional and Psychological Function - EQ-5D-5L | Week 0
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 1 and the highest possible score is 5, and a higher score indicates a worse outcome.
Emotional and Psychological Function - EQ-5D-5L | Week 2
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 1 and the highest possible score is 5, and a higher score indicates a worse outcome.
Emotional and Psychological Function - EQ-5D-5L | Week 6
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 1 and the highest possible score is 5, and a higher score indicates a worse outcome.
Emotional and Psychological Function - EQ-5D-5L | Week 12
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 1 and the highest possible score is 5, and a higher score indicates a worse outcome.
Quality of Life - EQ-5D-5L | Week -2
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 1 and the highest possible score is 5, and a higher score indicates a worse outcome.
Quality of Life - EQ-5D-5L | Week 0
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 1 and the highest possible score is 5, and a higher score indicates a worse outcome.
Quality of Life - EQ-5D-5L | Week 2
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 1 and the highest possible score is 5, and a higher score indicates a worse outcome.
Quality of Life - EQ-5D-5L | Week 6
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 1 and the highest possible score is 5, and a higher score indicates a worse outcome.
Quality of Life - EQ-5D-5L | Week 12
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 1 and the highest possible score is 5, and a higher score indicates a worse outcome.
Total Score - EQ-5D-5L | Week -2
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 5 and the highest possible score is 25, and a higher score indicates a worse outcome.
Total Score - EQ-5D-5L | Week 0
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 5 and the highest possible score is 25, and a higher score indicates a worse outcome.
Total Score - EQ-5D-5L | Week 2
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 5 and the highest possible score is 25, and a higher score indicates a worse outcome.
Total Score - EQ-5D-5L | Week 6
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 5 and the highest possible score is 25, and a higher score indicates a worse outcome.
Total Score - EQ-5D-5L | Week 12
  These outcomes will allow us to better understand the holistic effect of the intervention. The lowest possible score is 5 and the highest possible score is 25, and a higher score indicates a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Campbell, MD, Principal Investigator — Elisabeth Bruyere Hospital and The Ottawa Hospital
Locations (2):
- Canada (2):
  - The Ottawa Hospital, Ottawa, Ontario
  - Elisabeth Bruyere Hospital, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No